CLINICAL TRIAL: NCT05158868
Title: Effect of Post Covid-19 Hypoxia on Placenta of Normal Pregnant Women: A Possible Role of Hypoxia Inducible Factor-1α.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, FYAli, Principal investigator, Assiut University
Other Study IDs: Hif-1cov
Record Dates: First submitted 2021-12-14; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Hif-1α Covid-19
Keywords: Hif-1α covid-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post covid infected group: normal pregnant women infected by covid during 3rd trimester
  Interventions: Diagnostic Test: HiF-1 alpha measurement
- Control group: normal pregnant women
  Interventions: Diagnostic Test: HiF-1 alpha measurement

INTERVENTIONS:
Diagnostic Test: HiF-1 alpha measurement — HIF1- α is a heterodimeric transcription factor that bind to hypoxia response elements, which participates through the regulation of the expression of several genes in numerous cellular events such as O2 sensing, glucose metabolism, lipid metabolism, angiogenesis and other aspects of endothelial biology

SUMMARY:
To study the risk of hypoxia in placenta of normal pregnant women infected with covid-19 during third trimester of pregnancy.

DETAILED DESCRIPTION:
Hypoxaemia is an ominous sign of COVID-19, and it is usually an indicator of disease severity. An oxygen saturation above 90% is associated with better outcomes. Hypoxia indicates an imbalance of oxygen delivery to tissues and leads to compromised function.

The hypoxia-inducible factors (HIF) are considered master regulators of oxygen homeostasis and are oxygen level sensitive. HIF1a is a heterodimeric transcription factor that bind to hypoxia response elements, which participates through the regulation of the expression of several genes in numerous cellular events such as O2 sensing, glucose metabolism, lipid metabolism, angiogenesis and other aspects of endothelial biology.

PIGF is a proangiogenic protein and member of the vascular endothelial growth factor (VEGF) family. It is one of the key molecules in angiogenesis and vasculogenesis especially during embryogenesis and placental trophoblast is the main source of PIGF throughout the gestational period of pregnancy. It shares structural as well as amino acid sequence similarity with VEGF, but PIGF has binding afﬁnity only for VEGF receptor1(VEGFR-1). The inter-and intramolecular cross-talk between the VEGFR-1 and VEGFR-2 is regulated by PIGF. It binds toVEGFR-1 and displaces VEGF from this receptor, which results in activation and intermolecular trans phosphorylation of VEGFR-2 thereby amplify the VEGF-induced angiogenesis.

Hypoxic environment is essential for the proliferation and differentiation of cytotrophoblast for maintenance of materno-fetal circulation at early periods of pregnancy. But its prevalence in later stages of pregnancy causes several complications that may lead to maternal and fetal morbidity and mortality.

Several researchers have proved that the overexpression of HIF-1α is associated with the increased maternal serum concentration of soluble Fms-like tyrosine kinase 1 (sFlt1) during hypoxic conditions. High circulating levels of sFlt1 exerts an antiangiogenic state that is associated with low levels of proangiogenic factors, such as PIGF, and inhibition of PIGF with its receptor VEGFR-1.

Currently, there is no information regarding the expression of HIF-1a in normal pregnant women with COVID-19 infection and its potential involvement in the placentation of this condition. Therefore, in the present work we will detect the expression of hypoxia induced factor 1a (HIF1a) and possible molecular link between the expression of HIF-1α and PIGF based on previous studies which show significant negative association between HIF-1α and PIGF expression in patients suffering from preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* * Pregnant women who come for termination of pregnancy by CS or vaginal delivery

  * Gestational age is between 28-40 weeks.

The women will be divided into two groups:

* Covid-19 infection during 3rd trimester group (n = 25)
* Control normal pregnancy group (n = 25).

Exclusion Criteria:

* 1) Diabetes mellitus 2) Chronic hypertension 3) Preeclampsia 4) Acute or chronic infectious diseases or other chronic illness 5) Twins pregnancy 6) Anti phospholipid antibody syndrome

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: * Pregnant women who come for termination of pregnancy by CS or vaginal delivery
  * Gestational age is between 28-40 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The mean difference between HIF-1 between study groups | 1 week
  real time PCR and Immunohistochemistery of Hif-1α

REFERENCES:
- [Background] Young BE, Ong SWX, Kalimuddin S, Low JG, Tan SY, Loh J, Ng OT, Marimuthu K, Ang LW, Mak TM, Lau SK, Anderson DE, Chan KS, Tan TY, Ng TY, Cui L, Said Z, Kurupatham L, Chen MI, Chan M, Vasoo S, Wang LF, Tan BH, Lin RTP, Lee VJM, Leo YS, Lye DC; Singapore 2019 Novel Coronavirus Outbreak Research Team. Epidemiologic Features and Clinical Course of Patients Infected With SARS-CoV-2 in Singapore. JAMA. 2020 Apr 21;323(15):1488-1494. doi: 10.1001/jama.2020.3204. PMID 32125362
- [Background] Kashani KB. Hypoxia in COVID-19: Sign of Severity or Cause for Poor Outcomes. Mayo Clin Proc. 2020 Jun;95(6):1094-1096. doi: 10.1016/j.mayocp.2020.04.021. Epub 2020 Apr 23. No abstract available. PMID 32498766
- [Background] Majmundar AJ, Wong WJ, Simon MC. Hypoxia-inducible factors and the response to hypoxic stress. Mol Cell. 2010 Oct 22;40(2):294-309. doi: 10.1016/j.molcel.2010.09.022. PMID 20965423
- [Background] Iyer S, Leonidas DD, Swaminathan GJ, Maglione D, Battisti M, Tucci M, Persico MG, Acharya KR. The crystal structure of human placenta growth factor-1 (PlGF-1), an angiogenic protein, at 2.0 A resolution. J Biol Chem. 2001 Apr 13;276(15):12153-61. doi: 10.1074/jbc.M008055200. Epub 2000 Nov 7. PMID 11069911
- [Background] Autiero M, Waltenberger J, Communi D, Kranz A, Moons L, Lambrechts D, Kroll J, Plaisance S, De Mol M, Bono F, Kliche S, Fellbrich G, Ballmer-Hofer K, Maglione D, Mayr-Beyrle U, Dewerchin M, Dombrowski S, Stanimirovic D, Van Hummelen P, Dehio C, Hicklin DJ, Persico G, Herbert JM, Communi D, Shibuya M, Collen D, Conway EM, Carmeliet P. Role of PlGF in the intra- and intermolecular cross talk between the VEGF receptors Flt1 and Flk1. Nat Med. 2003 Jul;9(7):936-43. doi: 10.1038/nm884. PMID 12796773
- [Background] FOX H. THE VILLOUS CYTOTROPHOBLAST AS AN INDEX OF PLACENTAL ISCHAEMIA. J Obstet Gynaecol Br Commonw. 1964 Dec;71:885-93. doi: 10.1111/j.1471-0528.1964.tb04375.x. No abstract available. PMID 14243207
- [Background] Kingdom JC, Kaufmann P. Oxygen and placental villous development: origins of fetal hypoxia. Placenta. 1997 Nov;18(8):613-21; discussion 623-6. doi: 10.1016/s0143-4004(97)90000-x. PMID 9364596
- [Background] Nevo O, Soleymanlou N, Wu Y, Xu J, Kingdom J, Many A, Zamudio S, Caniggia I. Increased expression of sFlt-1 in in vivo and in vitro models of human placental hypoxia is mediated by HIF-1. Am J Physiol Regul Integr Comp Physiol. 2006 Oct;291(4):R1085-93. doi: 10.1152/ajpregu.00794.2005. Epub 2006 Apr 20. PMID 16627691
- [Background] Li H, Gu B, Zhang Y, Lewis DF, Wang Y. Hypoxia-induced increase in soluble Flt-1 production correlates with enhanced oxidative stress in trophoblast cells from the human placenta. Placenta. 2005 Feb-Mar;26(2-3):210-7. doi: 10.1016/j.placenta.2004.05.004. PMID 15708122